CLINICAL TRIAL: NCT04083157
Title: Intra-dermal With Topical Imiquimod Pretreatment Versus Intra-muscular Hepatitis B Vaccination in IBD Patients - a Double-blind Randomized Controlled Trial
Brief Title: Intra-dermal With Topical Imiquimod Pretreatment Versus Intra-muscular Hepatitis B Vaccination in IBD Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IBDHepBVaccine
Record Dates: First submitted 2019-09-02; First posted 2019-09-10 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Inflammatory Bowel Diseases; Hepatitis B
MeSH Terms: conditions — Inflammatory Bowel Diseases; Hepatitis B | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradermal hepatitis B vaccine with imiquimod (Experimental): Subjects in the study arm will receive 20 mcg intradermal Engerix-B at two separate sites (10 mcg/0.5 ml) with topical imiquimod ointment pre-treatment 5 minutes before injection.
  Interventions: Biological: Intradermal hepatitis B vaccine with imiquimod
- Intramuscular hepatitis B vaccine with aqueous cream (Active Comparator): Subjects in the control arm will receive 20 mcg intramuscular Engerix-B at two separate sites (10 mcg/ 0.5 ml) with topical placebo aqueous cream pretreatment 5 minutes before injection.
  Interventions: Biological: Intramuscular hepatitis B vaccine with aqueous cream

INTERVENTIONS:
Biological: Intradermal hepatitis B vaccine with imiquimod — Intradermal hepatitis B vaccine with topical imiquimod pretreatment
  Arms: Intradermal hepatitis B vaccine with imiquimod
Biological: Intramuscular hepatitis B vaccine with aqueous cream — Intramuscular hepatitis B vaccine with topical aqueous cream pretreatment
  Arms: Intramuscular hepatitis B vaccine with aqueous cream

SUMMARY:
Inflammatory bowel disease (IBD) has witnessed a rising incidence globally and in Hong Kong, an area where chronic hepatitis B (CHB) remains endemic. IBD patients are usually immunocompromised due to the disease itself and secondary to the use of medications including immunosuppressants and biologics, predisposing them to various opportunistic infection including hepatitis. Vaccination against hepatitis B virus (HBV) is recommended to prevent CHB and its related complications including flare up of acute hepatitis, cirrhosis and hepatocellular carcinoma. However, it is reported that efficacy with conventional intramuscular hepatitis B vaccination in IBD patients is suboptimal, especially among those receiving biologic therapies. Various strategies in boosting vaccine immunogenicity including the utilization of higher vaccination dose, shorter dosing interval, or alternate route of vaccine administration have been studied.6

Intradermal route of vaccination has been recently shown to be an effective way in augmenting immune response in specific patient groups who are known poor responders, including elderly and immunocompromised patients. In addition, topical imiquimod, a synthetic agonist of toll-like receptor 7 (TLR7), has been shown to further boost up the immunogenicity response when applied to the site before intradermal vaccination. The proposed study is the first clinical trial comparing the efficacy of intradermal hepatitis B vaccination with adjuvant topical application of imiquimod cream with the conventional intramuscular hepatitis B vaccination in IBD patients.

DETAILED DESCRIPTION:
Aim of study To compare the efficacy of intradermal hepatitis B vaccination with adjuvant topical imiquimod with conventional intramuscular hepatitis B vaccination in IBD patients.

Methodology Patient recruitment IBD patients newly referred to or currently followed up at Department of Medicine, Queen Mary Hospital will be screened for CHB status (HBsAg/Anti-HBs/Anti-HBc). Patients without CHB infection and evidence of prior HBV vaccination i.e. HBsAg -ve /Anti-HBc-ve/ Anti-HBs -ve will be recruited into the study. Eligible patients will be randomized to receive either intradermal vaccination with Engerix B with topical imiquimod or intramuscular vaccination with Engerix-B with topical aqueous cream as the control arm.

Randomization Eligible patients will be randomized in 1:1 ratio to receive intradermal hepatitis B vaccination (Engerix B) with topical imiquimod cream (as the study arm) or intramuscular hepatitis B vaccination (Engerix-B) with topical aqueous cream (as the control arm). Computer generated random number is used for randomization. Randomization sequences will be kept in opaque envelope and kept by a research staff not directly involved in this study. Once the patient has consented to the study, that research staff will open the envelope and notified the study nurse only of the vaccine allocation. In case of medical emergency or severe adverse reaction to the study medication, unblinding can be performed after notification of the principal investigator who will break the randomization code by revealing the randomization sequence assigned to the concerned study subject.

Vaccine administration Vaccination schedule is identical between the two arms with 3 doses given at 0, 1, 6 month. Participants in the study arm will receive 20 mcg intradermal Engerix-B at two separate sites (10 mcg/0.5 ml) with topical imiquimod ointment pre-treatment 5 minutes before injection. Participants in the control arm will receive 20 mcg intramuscular Engerix-B at two separate sites (10 mcg/ 0.5 ml) with topical placebo aqueous cream pretreatment 5 minutes before injection. The topical treatment will be given in a 4x4cm2 marked at the deltoid on each arm. Vaccination will be administered at clinic by dedicated study nurse, who is not involved in subsequent management of the participants. Both the investigators and the participants will be blinded to the result of randomization as only the study nurse know the route of administration.

Follow up Follow up visits will be arranged at 1,6,12 month after first dose of vaccine. Blood will be taken during each follow up visits for anti-HBs titres.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18 years old
* Confirmed IBD diagnosis (Ulcerative colitis, Crohns disease or IBD-Unclassified)
* HBsAg -ve / anti-HBs / antiHBc -ve
* Subjects must give written informed consent
* Subjects must be available to complete the study and comply with study procedures

Exclusion Criteria:

* Inability or unwilling to follow all required study procedures
* History of allergy or severe adverse reaction to the study vaccines, their components, topical imiquimod or aqueous cream
* Pregnant or lactating women
* HBsAg / anti-HBs / anti-HBc +ve
* Confirmed hepatitis C virus (HCV) (anti-HCV +ve) infection
* Fever (axillary temperature ≥ 38°C or oral temperature ≥ 38.5°C within 3 days of intended study vaccination, subjects can be recruited after the febrile episode subsides
* Have an active neoplastic disease
* Have any condition which the investigator believes may prevent successful completion of the study or interfere with results of the study
* Received an experimental agent (vaccine, drug, biologic, medication) within 1 month prior to vaccination or expect to receive an experimental agent during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Sero-protection rate to HBV | 12 months after first dose of vaccine
  Percentage of recruited subjects with anti-HBs titre ≥ 10 IU/L

SECONDARY OUTCOMES:
Injection site adverse effect of intradermal hepatitis B vaccine in IBD patients | up to 7 days after each dose of vaccination
  Injection site adverse effect recorded as following, with left and right arm recorded separately:
  Pain - 0 = no pain / 1 = pain on touch / 2 = pain during arm raising / 3 = pain on arm movement Presence or absence of the following Itching Swelling Hot sensation Bruise
Systemic adverse effect of intradermal hepatitis B vaccine in IBD patients | up to 7 days after each dose of vaccination
  Presence of absence of systemic adverse effect recorded as following:
  Fever Malaise Headache Myalgia Arthralgia Nausea Diarrhoea
Sero-protection rate to HBV at 1 and 6 months after dose of vaccine | 1 and 6 month after first dose of vaccine
Percentage of good responder defined as anti-HBs ≥ 100 IU/L | 12 month after first dose of vaccine
Geometric mean concentration of anti-HBs at 1, 6 and 12 months after first dose of vaccine | 1, 6 and 12 month after first dose of vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Wai Keung Leung, MD, Study Director — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ko KL, Lam YF, Cheung KS, Hung IF, Leung WK. Clinical trial: intra dermal hepatitis B vaccination with topical imiquimod versus intra muscular hepatitis B vaccination in patients with inflammatory bowel disease. Aliment Pharmacol Ther. 2022 Jul;56(2):301-309. doi: 10.1111/apt.16970. Epub 2022 May 11. PMID 35546255